CLINICAL TRIAL: NCT01156584
Title: A Phase 1 Ascending Dose Trial of the Safety and Tolerability of Toca 511 in Patients With Recurrent High Grade Glioma
Brief Title: A Study of a Retroviral Replicating Vector Combined With a Prodrug Administered to Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-08-01
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: glioma; glioblastoma; glioblastoma multiforme; Grade IV astrocytoma; brain cancer; recurrent glioblastoma; GBM; AA; AOD; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic oligoastrocytoma; malignant glioma; high grade glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — Genetic Therapy; Genetic Engineering; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Toca 511 vector/ Toca FC prodrug
  Interventions: Biological: Toca 511 vector; Drug: Toca FC

INTERVENTIONS:
Biological: Toca 511 vector — Single, stereotactic, transcranial, intratumoral injection or intravenous injection
  Other Names: Retroviral Replicating Vector (RRV); Gene Therapy; Gene Transfer
Drug: Toca FC — 4-6 week cycles of Toca FC. Doses evaluated from 120 mg/kg/day or 300 mg/kg/day. Duration of dosing evaluated: 6 days, 7 days or 14 days.
  Other Names: flucytosine, 5-FC, 5-FC XR, Toca FC (extended release flucytosine)

SUMMARY:
This is a multicenter, open-label, ascending-dose trial of the safety and tolerability of increasing doses of Toca 511, a Retroviral Replicating Vector (RRV), administered to patients with recurrent high grade glioma (rHGG) who have undergone surgery followed by adjuvant radiation therapy and chemotherapy. Patients will receive Toca 511 either via stereotactic, transcranial injection into their tumor or as an intravenous injection given daily for 3 & 5 days, depending on cohort. Approximately 3-4 weeks following injection of the RRV, treatment with Toca FC, an antifungal agent, will commence and will be repeated approximately every 6 weeks until study completion. After completion of this study, all patients will be eligible for enrollment and encouraged to enter a long-term continuation protocol that enables additional Toca FC treatment cycles to be given, as well as permits the collection of long-term safety and survival data.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* for intratumoral cohorts, supratentorial HGG (WHO grade III or IV)
* technically unresectable HGG
* initial definitive therapy such as surgery with or without adjuvant radiation
* subject elected not to undergo treatment with Gliadel wafer
* if receiving corticosteroids, dose is stable or decreasing for past 7 days
* KPS: at least 70
* absolute neutrophil count > 1500/mm^3
* absolute lymphocyte count > 500/mm^3
* platelet count > 100,000/mm^3
* hemoglobin > 10 g/dL
* for intratumoral cohort, coagulation profile favorable to surgery
* estimated glomerular filtration rate > 50 mL/min
* ALT < 3 times ULN and bilirubin < 1.5 mg/dL
* negative serum pregnancy test

Exclusion Criteria:

* cytotoxic therapy within the past 4 weeks (6 weeks for BCNU/CCNU)
* more than 2 recurrences including present recurrence
* Gliadel wafer or wafers implanted within the past 8 weeks
* taking more than 8 mg of dexamethasone per day
* for intratumoral cohorts, injection of tumor would require violation of ventricular system
* any infection requiring antibiotic, anticoagulant, or antiplatelet agents within the past 4 weeks
* for intratumoral cohort, bleeding diathesis or use of anticoagulants/antiplatelet agents that cannot be stopped
* allergy or intolerance to 5-FC
* HIV positive
* g.i. condition that would prevent ingestion or absorption of 5-FC
* any investigational treatment within the past 30 days
* pregnant or breast feeding
* received Avastin
* history of prior malignancy, excluding basal or squamous cell carcinoma of the skin, with an expected survival of less than 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-07; Primary Completion 2016-08-18 (Actual); Study Completion 2016-08-18 (Actual)

PRIMARY OUTCOMES:
Maximum Feasible, Safe and Well Tolerated Dose of Toca 511 | 8-10 weeks

SECONDARY OUTCOMES:
Safety and tolerability of repeated treatment with Toca FC following administration of Toca 511 | 6 months
  Review of adverse events including laboratory safety data (specifically any Grade 3 or higher non-hematologic toxicity or any Grade 4 or higher hematologic toxicity, felt to be related to Toca 511 or the Toca 511/Toca FC combination)
Overall survival of Subjects | Overall survivial, Overall survivial at 6 months (OS6), 9 months (OS9), and 12 months (OS12)
Evaluate progression free survival (PFS) at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asha Das, MD, Study Director — Tocagen Inc.; Manish Aghi, MD, NS, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - UCLA, Los Angeles, California
  - UCSD, San Diego, California
  - UCSF, San Francisco, California
  - Henry Ford Hospital, Detroit, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Methodist Hospital Research Institute, Houston, Texas

REFERENCES:
- [Background] Tai CK, Wang WJ, Chen TC, Kasahara N. Single-shot, multicycle suicide gene therapy by replication-competent retrovirus vectors achieves long-term survival benefit in experimental glioma. Mol Ther. 2005 Nov;12(5):842-51. doi: 10.1016/j.ymthe.2005.03.017. PMID 16257382
- [Background] Ostertag D, Amundson KK, Lopez Espinoza F, Martin B, Buckley T, Galvao da Silva AP, Lin AH, Valenta DT, Perez OD, Ibanez CE, Chen CI, Pettersson PL, Burnett R, Daublebsky V, Hlavaty J, Gunzburg W, Kasahara N, Gruber HE, Jolly DJ, Robbins JM. Brain tumor eradication and prolonged survival from intratumoral conversion of 5-fluorocytosine to 5-fluorouracil using a nonlytic retroviral replicating vector. Neuro Oncol. 2012 Feb;14(2):145-59. doi: 10.1093/neuonc/nor199. Epub 2011 Nov 9. PMID 22070930
- See also: Website for Accelerate Brain Cancer Cure — http://www.abc2.org
- See also: Website for the National Brain Tumor Society — http://www.braintumor.org